CLINICAL TRIAL: NCT01011361
Title: Red Cell Mass and Plasma Volume Measurements in Elderly Men and Women With Anemia
Status: Completed | Type: Observational
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Stanley L Schrier, Professor of Medicine (Hematology), Emeritus, Stanford University
Other Study IDs: IRB-16209; SU-07302009-3480 (Other: Stanford University)
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Last update posted 2016-03-24 (Estimated); Status verified 2016-03

CONDITIONS: Anemia
MeSH Terms: conditions — Anemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
On the basis that the clinical consequences of seemingly trivial levels of anemia are surprisingly severe, this study investigates if hemoglobin concentration accurately represents the underlying red cell mass in elderly patients with unresolved anemia.

DETAILED DESCRIPTION:
For the study, the routine clinical measurement of hemoglobin will be compared to true red cell mass and plasma volume in elderly patients with anemia.

ELIGIBILITY:
INCLUSION CRITERIA:

* 65 and older
* Anemia (hemoglobin < 13 g/dL in men or < 12 g/dL in women)
* Outpatient at either the Stanford Health Care (SHC) Medical Center or VA Palo Alto Health Care System

EXCLUSION CRITERIA:

* Body mass index (BMI):

  * < 18.5 kg/m2
  * > 35 kg/m2
* Palpable splenomegaly
* Contraindication to RBC mass/plasma volume testing
* On any experimental pharmacologic agent in the prior 2 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Outpatient elderly men and women (aged 65 years or older) with anemia, also enrolled in the "Anemia in the Elderly" NCT00640172 study.
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2009-04; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Red blood cell mass | 1 day

SECONDARY OUTCOMES:
Plasma volume measurements | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Stanley L Schrier, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No